CLINICAL TRIAL: NCT04921332
Title: Effect of Bright Light Therapy on Depression Symptoms in Adult Inpatients With Cystic Fibrosis (CF) and Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Bright Light Therapy for Depression Symptoms in Adults With Cystic Fibrosis (CF) and COPD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was stopped secondary to principal investigator needing to analyze data and present prior to graduating. Target enrollment not able to be reached prior to this.
Sponsor: Erica Osborn (Other)
Responsible Party: Sponsor-Investigator, Erica Osborn, Principal Investigator, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY20110407
Record Dates: First submitted 2021-06-02; First posted 2021-06-10 (Actual); Results first posted 2023-02-28 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Cystic Fibrosis; Depressive Symptoms; Chronic Obstructive Pulmonary Disease
Keywords: cystic fibrosis; depression; bright light therapy; adult; copd
MeSH Terms: conditions — Cystic Fibrosis; Depression; Pulmonary Disease, Chronic Obstructive | interventions — Ultraviolet Therapy

STUDY DESIGN:
Intervention Model Description: This is a non-randomized, single group, pre- and post-intervention project.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Bright Light Therapy (BLT) (Experimental): The intervention will consist of daily BLT sessions lasting 30 minutes at approximately 10AM (since many CF and COPD patients may not awaken until this time) starting on the day of admission through discharge for a goal of seven consecutive days. The intervention will use a 10,000-lux light box placed approximately 16-24 inches from the patient's face.
  Interventions: Device: Bright Light Therapy (BLT) Lamp

INTERVENTIONS:
Device: Bright Light Therapy (BLT) Lamp — With its built in automatic timer shut-off function, the bedside registered nurse (RN) would not need to return to the room to turn off this lamp after 30 minutes because the lamp will automatically shut off on its own.
  Other Names: Verilux HappyLight Luxe - UV-Free LED Therapy Lamp by Verilux

SUMMARY:
This is a project that will determine whether the use of daily bright light therapy has an effect on depressive symptoms experienced by adult inpatients with CF and COPD. The purpose of this project is to apply a daily 30-minute BLT intervention to hospitalized adult CF and COPD patients in order to decrease symptoms of depression as measured by depression inventory scoring.

DETAILED DESCRIPTION:
This project will occur on a 29-bed pulmonary step-down unit at a 1,600-bed academic medical center. This unit commonly treats patients with CF, COPD, and other pulmonary complications. The unit's patient care staff will be educated on the bright light lamps in order to prevent interruptions and to encourage compliance.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with cystic fibrosis or chronic obstructive pulmonary disease (COPD)
* Adult age 18 or older
* Admitted to the pulmonary step-down and transplant unit
* Score greater than zero on pre-intervention Beck's Depression Inventory-II (BDI-II)

Exclusion Criteria:

* Pre-existing ophthalmological conditions or photosensitivity
* Migraines
* Receiving high dose steroids for transplant rejection (due to mood altering qualities),
* Antibiotics that increase light sensitivity
* Diagnosed with bipolar disorder (light therapy may trigger mania)
* Admissions anticipated to span less than 48 hours
* Children are being excluded due to the fact that only adult CF and COPD subjects are admitted to University of Pittsburgh Medical Center (UPMC) Presbyterian hospital

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2021-09-07 (Actual); Primary Completion 2022-03-22 (Actual); Study Completion 2022-03-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erica Osborn, BSN, Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - University of Pittsburgh Medical Center Presbyterian Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Data produced from this project may be shared with investigators conducting research on a similar topic within the University of Pittsburgh and outside. Shared information from this project will be de-identified under an approved DUA.
Supporting Information: CSR
Time Frame: Results and data from this study will be available immediately and maintained for seven years following completion.
Access Criteria: Investigators conducting research on a similar topic within the University of Pittsburgh and outside

REFERENCES:
- [Background] Kopp BT, Hayes D Jr, Ghera P, Patel A, Kirkby S, Kowatch RA, Splaingard M. Pilot trial of light therapy for depression in hospitalized patients with cystic fibrosis. J Affect Disord. 2016 Jan 1;189:164-8. doi: 10.1016/j.jad.2015.08.056. Epub 2015 Sep 28. PMID 26433764
- [Background] Guzel Ozdemir P, Boysan M, Smolensky MH, Selvi Y, Aydin A, Yilmaz E. Comparison of venlafaxine alone versus venlafaxine plus bright light therapy combination for severe major depressive disorder. J Clin Psychiatry. 2015 May;76(5):e645-54. doi: 10.4088/JCP.14m09376. PMID 26035199
- [Background] Lam RW, Levitt AJ, Levitan RD, Michalak EE, Cheung AH, Morehouse R, Ramasubbu R, Yatham LN, Tam EM. Efficacy of Bright Light Treatment, Fluoxetine, and the Combination in Patients With Nonseasonal Major Depressive Disorder: A Randomized Clinical Trial. JAMA Psychiatry. 2016 Jan;73(1):56-63. doi: 10.1001/jamapsychiatry.2015.2235. PMID 26580307

RESULTS

PARTICIPANT FLOW:
Groups:
- Bright Light Therapy (BLT): The intervention will consist of daily BLT sessions lasting 30 minutes at approximately 10AM (since many CF and COPD patients may not awaken until this time) starting on the day of admission through discharge for a goal of seven consecutive days. The intervention will use a 10,000-lux light box placed approximately 16-24 inches from the patient's face.
  Bright Light Therapy (BLT) Lamp: With its built in automatic timer shut-off function, the bedside RN would not need to return to the room to turn off this lamp after 30 minutes because the lamp will automatically shut off on its own.
Period: Overall Study
Arm/Group | Bright Light Therapy (BLT)
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Bright Light Therapy (BLT)
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.25 (20.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 4
Diagnosis [Count of Participants; unit: Participants]
  Cystic Fibrosis | 3
  Chronic Obstructive Pulmonary Disease | 1
Pre-intervention BDI-II Scoring [Mean (Standard Deviation); unit: Score on a scale] — Self-reported answer total to the 21 scored items on BDI-II (minimum score obtainable=0 (absent symptoms); maximum score obtainable=63 (most severe symptoms). Higher score=worse outcome.
  Score on a scale | 24.75 (8.995)

OUTCOME MEASURES:

1. Primary Outcome: Change in Pre- and Post-intervention Beck's Depression Inventory II Scores (BDI-II)
Description: Change between pre-intervention and post-intervention self-reported answer totals to the 21 scored items on BDI-II (minimum score obtainable=0 (absent symptoms); maximum score obtainable=63 (most severe symptoms).
Time Frame: First at time of admission, second at end of 7 day goal or upon discharge.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bright Light Therapy (BLT)
Number analyzed (Participants) | 4
score on a scale | 8.750 (10.63)

2. Secondary Outcome: Number of Days Until Completion of Daily Bright Light Therapy (BLT)
Description: The RN will sign a daily log indicating what time therapy was initiated and if therapy was refused. These logs will be collected from patient doors at the end of each week by the principal investigator (PI) in order to measure compliance with completion of therapy on a daily basis.
Time Frame: Daily for duration of intervention period (goal/maximum of 7 days).
Measure: Mean (Standard Deviation); unit: days
Groups:
- Bright Light Therapy Compliance (Secondary Outcome): The RN will sign a daily log indicating what time therapy was initiated and if therapy was refused. These logs will be collected from patient doors at the end of each week by the principal investigator (PI) in order to measure compliance with completion of therapy on a daily basis.
Arm/Group | Bright Light Therapy Compliance (Secondary Outcome)
Number analyzed (Participants) | 4
days | 4.5 (5)

ADVERSE EVENTS:
Time Frame: Adverse events were monitored for and collected over the implementation period of this study which spanned over 7 months.
Arm/Group | Bright Light Therapy (BLT)
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

LIMITATIONS AND CAVEATS:
Limitations include a smaller than needed sample size to reach statistically reliable results, inconsistency with daily compliance among participants, limited nursing staff availability, potential bias (patient's knew the purpose of the study, this was not blind), lack of generalizability (e.g. risk of participant bias, single site location, situational factors, working with specialty population), and factors surrounding completion of this study during the COVID-19 pandemic.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-03-30): https://cdn.clinicaltrials.gov/large-docs/32/NCT04921332/Prot_SAP_000.pdf
  • Informed Consent Form (2021-12-28): https://cdn.clinicaltrials.gov/large-docs/32/NCT04921332/ICF_002.pdf